CLINICAL TRIAL: NCT02161367
Title: A Randomized Controlled Trial of the Effect of Simethicone on Postoperative Ileus in Patients Undergoing Colorectal Surgery: A Pilot Study
Brief Title: Effect of Simethicone on Postoperative Ileus in Patients Undergoing Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simethicone-CRSurgery-1415
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Ileus; Ileus
Keywords: colorectal surgery; postoperative ileus; simethicone; randomized controlled trial; double blind; pilot study; anti-foaming agent; abdominal pain; abdominal distention; nausea vomiting; flatus; bowel movement; placebo; postoperative complications; polydimethylsiloxane; hydrated silica gel; gas bubbles; intestinal tract
MeSH Terms: conditions — Ileus; Abdominal Pain; Flatulence; Postoperative Complications | interventions — Simethicone; Excipients

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Simethicone, OVOL (Experimental): Patients in the intervention arm will receive, in a blinded fashion, 160mg of simethicone orally four times a day for the first five postoperative days. Patients will be evaluated by a trained research assistant on a daily basis while in hospital. Passage of flatus, bowel movements, and postoperative pain will be evaluated at those visits. A two-week, and 30-day phone call to patients discharged from hospital will be done to assess for outcomes after discharge. Follow-up will end after the 30th postoperative day.
  Interventions: Drug: Simethicone
- Oral Suspending Vehicle, Ora-Plus (Placebo Comparator): Patients in the control arm will receive, in a blinded fashion, 160mg of the placebo orally four times a day for the first five postoperative days. The placebo will be prepared by pharmacy to be identical to the test drug formulation except for being pharmacologically inert. Patients will be evaluated by a trained research assistant on a daily basis while in hospital. Passage of flatus, bowel movements, and postoperative pain will be evaluated at those visits. A two-week, and 30-day phone call to patients discharged from hospital will be done to assess for outcomes after discharge. Follow-up will end after the 30th postoperative day.
  Interventions: Drug: Oral Suspending Vehicle

INTERVENTIONS:
Drug: Simethicone — Pharmacological category: antiflatulent
  160mg Simethicone orally, 4 times a day for the first five postoperative days
  Other Names: OVOL®
  Arms: Simethicone, OVOL
Drug: Oral Suspending Vehicle — ORA-Plus is an aqueous-based vehicle.
  Identical to the test drug formulation except for being pharmacologically inert. 160mg Ora-Plus orally, 4 times a day for the first five postoperative days
  Other Names: ORA-Plus®
  Arms: Oral Suspending Vehicle, Ora-Plus

SUMMARY:
Post-operative ileus is a common complication following abdominal surgery. It results in abdominal distension, nausea and vomiting as well as abdominal pain. Furthermore, this results in prolonged hospital stay and occasionally readmission following abdominal surgery.The etiology of post-operative ileus is multifactorial and studies evaluating potential treatment options are abundant, though few reliable interventions exist. This study proposal describes a double-blinded randomized controlled trial investigating the effect of simethicone on post-operative ileus in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Simethicone is an orally administered anti-foaming agent comprised of polydimethylsiloxane and hydrated silica gel. Its leads to the coalescence of gas bubbles in the intestinal tract, facilitating its emission. To date, there are no contemporary studies evaluating the efficacy of simethicone on POI in patients undergoing colorectal surgery.

The proposed study is a pilot double-blinded randomized controlled trial of simethicone versus placebo in patients undergoing colorectal surgery. Starting on postoperative day one, patients in the experimental arm of the study will receive, in a blinded fashion, 160mg of simethicone orally four times a day for the first five postoperative days. Patients assigned to the control arm will receive a placebo agent orally with the same frequency and duration.

All consenting patients over the age of 18 undergoing elective, abdominal colorectal surgery involving bowel resection with or without re-anastomosis at either the Juravinski Hospital and Cancer Center or St. Joseph's Hospital in Hamilton, Ontario will be enrolled. This will include patients undergoing both open and laparoscopic surgery.

Patients will be prospectively evaluated by a trained research assistant on a daily basis while in hospital. Passage of flatus, bowel movements, and postoperative pain will be evaluated at those visits. A two-week, and 30-day phone call to patients discharged from hospital will be done to assess for outcomes after discharge. Follow-up will end after the 30th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients over the age of 18 undergoing elective, abdominal colorectal surgery involving bowel resection with or without re-anastomosis (both open and laparoscopic surgeries) at either the Juravinski Hospital and Cancer Center or St. Joseph's Hospital in Hamilton

Exclusion Criteria:

* Patients undergoing emergency surgery
* Documented allergy to simethicone
* Unable to provide informed consent (non-English speaking patients and those with cognitive impairment)
* Patients not having an abdominal operation (ie. perineal procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
time to first passage of flatus | participants will be followed for the duration of their hospital stay, an expected average of 7 days
  passage of flatus (measured in hours) is considered an acceptable sign of the return of gut function and a criterion for discharge from hospital (bowel movement is not)

SECONDARY OUTCOMES:
time to first bowel movement | participants will be followed for the duration of their hospital stay, an expected average of 7 days
length of hospital stay | participants will be followed for the duration of their hospital stay, an expected average of 7 days
postoperative pain | participants will be followed for the duration of their hospital stay, an expected average of 7 days
  measured using the Visual Analogue Scale for pain
postoperative narcotic requirements | participants will be followed for the duration of their hospital stay, an expected average of 7 days
incidence of postoperative vomiting | participants will be followed for the duration of their hospital stay, an expected average of 7 days
incidence of postoperative complications | within the first 30 days (plus or minus 3 days) after surgery
  including but not limited to wound and anastomotic occurences, bleeding, infections, readmission to hospital, death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn S Forbes, MD, MSc, Principal Investigator — McMaster University; Cagla Eskicioglu, MD, MSc, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

REFERENCES:
- [Background] Doorly MG, Senagore AJ. Pathogenesis and clinical and economic consequences of postoperative ileus. Surg Clin North Am. 2012 Apr;92(2):259-72, viii. doi: 10.1016/j.suc.2012.01.010. PMID 22414412
- [Background] Story SK, Chamberlain RS. A comprehensive review of evidence-based strategies to prevent and treat postoperative ileus. Dig Surg. 2009;26(4):265-75. doi: 10.1159/000227765. Epub 2009 Jul 3. PMID 19590205
- [Background] Kehlet H, Holte K. Review of postoperative ileus. Am J Surg. 2001 Nov;182(5A Suppl):3S-10S. doi: 10.1016/s0002-9610(01)00781-4. PMID 11755891
- [Background] Senagore AJ. Pathogenesis and clinical and economic consequences of postoperative ileus. Am J Health Syst Pharm. 2007 Oct 15;64(20 Suppl 13):S3-7. doi: 10.2146/ajhp070428. PMID 17909274
- [Background] Barletta JF, Asgeirsson T, Senagore AJ. Influence of intravenous opioid dose on postoperative ileus. Ann Pharmacother. 2011 Jul;45(7-8):916-23. doi: 10.1345/aph.1Q041. Epub 2011 Jul 5. PMID 21730280
- [Background] Sternini C, Patierno S, Selmer IS, Kirchgessner A. The opioid system in the gastrointestinal tract. Neurogastroenterol Motil. 2004 Oct;16 Suppl 2:3-16. doi: 10.1111/j.1743-3150.2004.00553.x. PMID 15357847
- [Background] Bauer AJ, Boeckxstaens GE. Mechanisms of postoperative ileus. Neurogastroenterol Motil. 2004 Oct;16 Suppl 2:54-60. doi: 10.1111/j.1743-3150.2004.00558.x. PMID 15357852
- [Background] Hocevar BJ, Robinson B, Gray M. Does chewing gum shorten the duration of postoperative ileus in patients undergoing abdominal surgery and creation of a stoma? J Wound Ostomy Continence Nurs. 2010 Mar-Apr;37(2):140-6. doi: 10.1097/WON.0b013e3181d0b92b. PMID 20228654
- [Background] Danhof IE, Stavola JJ. Accelerated transit of intestinal gas with simethicone. Obstet Gynecol. 1974 Jul;44(1):148-54. No abstract available. PMID 4600627
- [Background] Gibstein A, Cooper JJ, Wisot AL, Rosenthal AH. Prevention of postoperative abdominal distention and discomfort with simethicone. Obstet Gynecol. 1971 Sep;38(3):386-90. No abstract available. PMID 4937581
- [Background] Chan MK, Law WL. Use of chewing gum in reducing postoperative ileus after elective colorectal resection: a systematic review. Dis Colon Rectum. 2007 Dec;50(12):2149-57. doi: 10.1007/s10350-007-9039-9. PMID 17710495
- [Background] Forbes SS, Stephen WJ, Harper WL, Loeb M, Smith R, Christoffersen EP, McLean RF. Implementation of evidence-based practices for surgical site infection prophylaxis: results of a pre- and postintervention study. J Am Coll Surg. 2008 Sep;207(3):336-41. doi: 10.1016/j.jamcollsurg.2008.03.014. Epub 2008 May 19. PMID 18722937
- [Background] Eskicioglu C, Gagliardi A, Fenech DS, Victor CJ, McLeod RS. Can a tailored knowledge translation strategy improve short term outcomes? A pilot study to increase compliance with bowel preparation recommendations in general surgery. Surgery. 2011 Jul;150(1):68-74. doi: 10.1016/j.surg.2011.02.010. Epub 2011 May 18. PMID 21596413